CLINICAL TRIAL: NCT06486155
Title: Evaluation of Axillary Lymph Node Metastasis Status of Breast Cancer Based on Pathological Images and Virtual Staining
Status: Not yet recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Collaborators: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: KYLX2024-129
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-06

CONDITIONS: Virtual Staining; Lymph Node Metastasis; Breast Cancer; Digital Pathology
MeSH Terms: conditions — Lymphatic Metastasis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop an artificial intelligence model to transform unstained lymph node tissue slice images directly into stained images. The main questions it aims to answer are:

Can the virtual staining model generate hematoxylin and eosin (H&E) and immunohistochemistry (IHC) images suitable for clinical diagnosis from unstained paraffin-embedded lymph node slice images, including those from breast axillary lymph nodes and other tumor lymph nodes?

Can the virtual staining model generate H&E and IHC images suitable for clinical diagnosis from unstained frozen sentinel lymph node slice images from breast cancer patients?

Researchers will retrospectively collect paraffin-embedded lymph node slices from tumor patients and prospectively collect frozen sentinel lymph node slices from breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

Female patients aged 18-75 with breast cancer; Undergoing surgical excision of breast cancer and sentinel lymph node biopsy/axillary lymph node dissection; Lymph nodes with clear postoperative paraffin pathological results.

Part 2:

Patients aged 18-75 with one of the following cancers: thyroid, lung, esophagus, stomach, colorectal, prostate, bladder, or cervix; Undergoing surgical resection of lymph nodes; Lymph nodes with clear postoperative paraffin pathological results.

Part 3:

Female patients aged 18-75 with breast cancer; Undergoing surgical excision of breast cancer and sentinel lymph node biopsy; Sentinel lymph nodes with clear postoperative paraffin pathological results.

Exclusion Criteria:

Part 1 / Part 2:

Lymph node diagnosis is missing; Absence of lymph node component in the slice.

Part 3:

Sentinel lymph node diagnosis is missing; Absence of lymph node component in the frozen slice.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part 1:
  The investigators plan to collect 1000 patients with breast cancer.
  Part 2:
  The investigators plan to collect 100 patients with each of the following cancers: thyroid, lung, esophagus, stomach, colorectal, prostate, bladder, and cervix. The total number of patients will be 800.
  Part 3:
  The investigators plan to prospectively collect 400 patients with breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lymph node metastasis status | 2024-2025
  Lymph node metastasis status: metastasis or non-metastasis
Accuracy, Sensitivity, Specificity，Area under the curve， | 2024-2025
  The performance of pathologists diagnosing the lymph node metastasis status by virtual and real staining whole slide images
Positive predictive value，Negative predictive value | 2024-2025
  The performance of pathologists diagnosing the lymph node metastasis status by virtual and real staining whole slide images

SECONDARY OUTCOMES:
Peak Signal-to-Noise Ratio(PSNR) | 2024-2025
  Scores of the similarity between virtual and real staining of lymph nodes, with values ranging from 0 to infinity, the higher scores mean the better outcomes
Multi-Scale Structural Similarity (MS-SSIM) | 2024-2025
  Scores of the similarity between virtual and real staining of lymph nodes, with values ranging from 0 to 1, the higher scores mean the better outcomes
Pearson correlation coefficient | 2024-2025
  Scores of the similarity between virtual and real staining of lymph nodes, with values ranging from 0 to 1, the higher scores mean the better outcomes